CLINICAL TRIAL: NCT05952232
Title: A Randomized, Double-blind, Placebo-controlled, Feasibility Study to Evaluate Efficacy of Different Natural Ingredients in Improving Gut Health in Adults With Leaky Gut - a Pilot Study
Brief Title: A Study to Evaluate Efficacy of Different Natural Ingredients in Improving Gut Health in Adults With Leaky Gut.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EB/230301/TPEKC/LG
Record Dates: First submitted 2023-06-22; First posted 2023-07-19 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Gut Health

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PA-GH-01 (Active Comparator): 1 capsule after breakfast once a day
  Interventions: Dietary Supplement: PA-GH-01
- MK-GH-04 (Active Comparator): 1 capsule after breakfast once a day
  Interventions: Dietary Supplement: MK-GH-04
- TSH-GH-03 (Active Comparator): 1 capsule after breakfast once a day
  Interventions: Dietary Supplement: TSH-GH-03
- PA-GH-02 (Placebo Comparator): 1 capsule after breakfast once a day
  Interventions: Dietary Supplement: PA-GH-02

INTERVENTIONS:
Dietary Supplement: PA-GH-01 — 1 capsule after breakfast once a day
  Arms: PA-GH-01
Dietary Supplement: MK-GH-04 — 1 capsule after breakfast once a day
  Arms: MK-GH-04
Dietary Supplement: TSH-GH-03 — 1 capsule after breakfast once a day
  Arms: TSH-GH-03
Dietary Supplement: PA-GH-02 — 1 capsule after breakfast once a day
  Arms: PA-GH-02

SUMMARY:
The present study is a randomized, placebo-controlled, double-blind, parallel group study to assess the gut health effects of IP as compared to a placebo in overweight individuals experiencing gut issues. Approximately 20 participants aged between 18 and 65 years will be screened for each group. All the five arms of the IP and placebo trial arms will each have at least 10 completed participants after accounting for the screening failure and dropout/withdrawal rate of 20% each. The treatment duration for all the study participants will be 29 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals with the age ≥18 and ≤65 years with moderate physical activity level as per International Physical Activity Questionnaire - Short Form (IPAQ-SF)
* Body mass index > 18 and < 29.9 kg/m2
* Individuals with at least once/ week complains of ≥ 3 of following gastrointestinal symptoms since last three months: dyspepsia, diarrhea, constipation, heartburn, nausea, acid reflux, bloating.
* Individuals agreeing to consume four tablets (325 mg each) of aspirin twice within a 12-hour period
* Individuals with fasting blood glucose levels ≤ 125 mg/dL
* Individuals with availability of western toilet at their homes for stool sample collection
* Individuals who are literate enough to understand the essence of study, are informed about the purpose of the study, and understand their rights.
* Individuals who are able to give written informed consent and are willing to participate in the study.

Exclusion Criteria:

* Individuals diagnosed with IBS including IBS-Constipation, IBS-Mixed, IBS-Diarrhea or Unclassified
* Allergy to aspirin
* Use of medications in the last 2 weeks prior to the pre-baseline period. This does not include birth control pills or standard multi-vitamin/mineral supplements
* Performing high intensity exercise regularly using IPAQ- SF
* Daily use of NSAIDs in the last 3 months or incidental use in the last 2 weeks prior to screening
* Unwillingness to avoid the use of antidiarrheal or laxative medication on a regular or an "as-needed basis" during the full length of the study
* Abnormal Thyroid Stimulating Hormone (TSH) value which is < 0.40 or > 4.50 μIU/mL
* Individuals with uncontrolled type II DM defined as FBG > 125 mg/ dL
* Presence of uncontrolled hypertension defined as SBP ≥ 140 mm Hg and/or DBP ≥ 90 mm Hg with or without anti-hypertensives
* Individuals on high-fiber/ fodmap diet
* Individuals with known diagnosis of helicobacter pylori infection
* Individuals with a history of surgical resection of the stomach, small intestine or large intestine
* Individuals with a history of or complications from inflammatory bowel disease (Crohn's disease or ulcerative colitis) and ischemic colitis
* Current smokers
* Use of another investigational product within 3 months of the screening visit
* History or current impaired cardiovascular circulation or uncontrolled hypertension, diabetes, bleeding tendencies, kidney, liver or chronic respiratory diseases including asthma, or any other disease, that by the investigators' discretion could interfere with the intestinal barrier function of the subject
* Individuals who used probiotics, prebiotics, antibiotics, prokinetics, laxatives, suppositories or enemas in the last 3 months
* Individuals with a history of any diet-based intolerance (gluten or lactose intolerance)
* Individuals with a history of or complications from malignant tumors.
* History of any significant neurological and psychiatric condition which may affect the participation and inference of the study's end points.
* Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine dependence.
* High-risk drinking as defined by consumption of 4 or more alcohol containing beverages on any day or 8 or more alcohol containing beverages per week for women and 5 or more alcohol containing beverages on any day or 15 or more alcohol containing beverages per week for men
* Individuals who have clinically significant following illness, i.e., Cardiovascular, endocrine system, immune system, respiratory system, hepatobiliary system, kidney and urinary system, neuropsychiatric, musculoskeletal, inflammatory, blood and tumors, other gastrointestinal diseases, etc
* Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives
* Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of the natural ingredients on gut permeability as assessed by the change in | Day 29
  Gut permeability as assessed by the urinary lactulose-mannitol ratio from baseline
To assess efficacy of the natural ingredients on gut permeability as assessed by the change in | Day 29
  Gut protection as assessed by the Aspirin challenge test from baseline
To assess efficacy of the natural ingredients on gut permeability as assessed by the change in | Day 29
  Stool consistency as assessed by Bristol Stool Type from baseline
To assess efficacy of the natural ingredients on gut permeability as assessed by the change in | Day 29
  Gut microbiome as assessed by the fecal pH from baseline
To assess efficacy of the natural ingredients on gut permeability as assessed by the change in | Day 29
  Quality of life as assessed by gastrointestinal quality of life index (GIQLI) from baseline
To assess efficacy of the natural ingredients on gut permeability as assessed by the change in | Day 29
  The stress level as assessed by change in the Perceived Stress Scale (PSS) from baseline
To assess efficacy of the natural ingredients on gut permeability as assessed by the change in | Day 29
  Appetite regulation as assessed by a Three-Factor Eating Questionnaire-R18 (TFEQ-R18) from baseline
To assess efficacy of the natural ingredients on gut permeability as assessed by the change in | Day 29
  Motivation to exercise as assessed by VAS score from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Dr. Kumta Mali's Clinic, Mumbai, Maharashtra
  - Dr. Preeti Bawaskar's Clinic, Thane, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided